CLINICAL TRIAL: NCT05708807
Title: FIND Stroke Recovery: A Longitudinal Frequent Evaluation Long-term Follow-up Study
Brief Title: FIND Stroke Recovery - A Longitudinal Study
Acronym: FIND
Status: Recruiting | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: FIND
Record Dates: First submitted 2022-12-21; First posted 2023-02-01 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Stroke Hemorrhagic; Stroke, Ischemic; Risk Factor, Cardiovascular; Cognitive Impairment
Keywords: recovery; rehabilitation; stroke severity; plasticity; modified Rankin Scale; National Institutes of Health Stroke Scale; Fugl-Meyer assessment; blood sampling; stroke subtype
MeSH Terms: conditions — Stroke; Hemorrhagic Stroke; Ischemic Stroke; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Protocol At admission participants undergo adequate neuroimaging and additional work-up according to clinical routine and answer questionaries on medical history, education, occupancy, pre-stroke functionality and donate blood samples. At 3 and 6 months and 1, 2 and 5 years the participants come for follow ups where they undergo substantial testing on cognition and motor function in parallel they also answer questionaries on mood, health, participation and recovery and donate blood samples. A detailed protocol will be published as a "study protocol".
  Biomarkers Blood samples are transferred to the Biobank West, Sahlgrenska University Hospital, Region Västra Götaland, where samples will be aliquoted and stored at -80 °C in a locked space, further details in the full study protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational - all: All included stroke patients.
  Interventions: Other: Observational - all

INTERVENTIONS:
Other: Observational - all — All stroke patients are included.

SUMMARY:
Stroke survivors frequently suffer disabilities including motor and cognitive problems, impairments in speech and vision, depression, and several other disabilities that worsen their quality of life. Some will recover fully after stroke and others will have permanent impairments. Few studies show trajectories of recovery in different domains after stroke, hence recovery time-lines are not fully known. Also, the whole range of mechanisms leading to recovery are not precisely known (1). To monitor those mechanisms one can utilize biomarkers.

In parallel to the studies of recovery, studies on time series of biomarkers after stroke are limited (2). Hence, a crucial first step to increase knowledge on biomarkers of stroke recovery is to gain a better understanding of the time course of both stroke recovery and biomarker patterns. Biomarkers can later be used for outcome predictions after stroke.

DETAILED DESCRIPTION:
BACKGROUND

Stroke survivors frequently suffer disabilities including motor and cognitive problems, impairments in speech and vision, depression, and several other disabilities that worsen their quality of life. Some will recover fully after stroke and others will have permanent impairements. Few studies show trajectories of recovery in different domains after stroke, hence recovery time-lines are not fully known. Also, the whole range of mechanisms leading to recovery are not precisely known (1). To monitor those mechanisms one can utilize biomarkers.

In parallel to the studies of recovery, studies on time series of biomarkers after stroke are limited (2). Hence, a crucial first step to increase knowledge on biomarkers of stroke recovery is to gain a better understanding of the time course of both stroke recovery and biomarker patterns. Biomarkers can later be used for outcome predictions after stroke.

WORK PLAN

AIM Determine temporal profiles describing the speed, order, and degree of recovery in neurological and cognitive functions in various domains with simultaneous profiling of changes in blood biomarker concentrations, in the acute, subacute phases and long-term of stroke. Determine individual and interindividual variations in recovery in the different domains.

Informed consent Written informed consent will be obtained from all willing participants or their next-of-kin.

ELIGIBILITY:
Investigators enrol patients presenting with first-ever ischemic stroke or intracerebral haemorrhage admitted to the stroke units at the Sahlgrenska University Hospital in Gothenburg, Sweden.

The inclusion criteria are:

• first-ever acute ischemic stroke; or intracerebral hemorrhage.

The exclusion criteria are:

* pre-stroke mRS score of ≥3;
* severe neurodegenerative disease, cerebral neoplasm or terminal illness; and
* patients considered unlikely to be able to participate in or to understand and/or comply with study procedures during follow-up visits at the hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators enrol patients presenting with first-ever ischemic stroke or intracerebral haemorrhage admitted to the stroke units at the Sahlgrenska University Hospital in Gothenburg, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Medical data Clinical data | Baseline, and change from baseline at 3, 6 and 12 months; 2 and 5 years.
  Stroke subtype, medical history, life style questions between baseline and follow-ups
Stroke severity | Baseline, and change from baseline at 3, 6 and 12 months; 2 and 5 years.
  Change of National Institutes of Health Stroke Scale (NIHSS) between baseline and follow-ups.
Functional independence | Pre-stroke estimation, baseline, and change from baseline at 3, 6 and 12 months; 2 and 5 years.
  Change of modified Ranking Scale (mRS) functional independence
Walking ability | Baseline, and change from baseline at 3, 6 and 12 months; 2 and 5 years.
  Change in functional Ambulation Category between baseline and follow ups.
Postural control | Baseline, and change from baseline at 3, 6 and 12 months; 2 and 5 years.
  Change in postural control, evaluated by Berg Balance Scale (BBS), between baseline and follow ups.
Blood samples | Baseline, and change from baseline at 3, 6 and 12 months; 2 and 5 years
  Analyses of plasma protein levels and circulating RNA profiles in comparison to baseline
FMA-arm test | Baseline, and change from baseline at 3, 6 and 12 months; 2 and 5 years
  Change in performance on Fugl-Meyer Assessment of Motor Recovery after Stroke test between baseline and follow-up.
SAFE | Baseline, and change from baseline at 3, 6 and 12 months; 2 and 5 years
  Change in performance on Shoulder Abduction and Finger Extension (SAFE) score between baseline and follow ups.
MoCA | Baseline, and change from baseline at 3, 6 and 12 months; 2 and 5 years
  Change in the Montreal Cognitive Assessment between baseline and follow ups.
Neuroimaging | Baseline, and change from baseline at 3, and 12 months; 2 years
  Changes in MRI scans between baseline and follow-ups.
D-FIS | Baseline, and change from baseline at 3, 6 and 12 months; 2 and 5 years
  Change in the Daily Fatigue Impact Scale (D-FIS) between baseline and follow ups.
HAD | Baseline, and change from baseline at 3, 6 and 12 months; 2 and 5 years
  Change in the Hospital Anxiety and Depression (HAD) scale between baseline and follow ups.
SIS | Baseline, and change from baseline and 3, 6 and 12 months; 2 and 5 years
  Change in domains of Stroke Impact Scale (SIS) between baseline and follow ups.
FAS | Baseline, and change from baseline at 3, 6 and 12 months; 2 and 5 years
  Change in the Verbal Fluency Test between baseline and follow ups.
CWT | Baseline, and change from baseline at 3, 6 and 12 months; 2 and 5 years
  Change in the Color-Word Interference test between baseline and follow ups.
TMT | Baseline, and change from baseline at 3, 6 and 12 months; 2 and 5 years
  Change in the Trail Making Test between baseline and follow ups.
RBANS | Baseline, and change from baseline at 3, 6 and 12 months; 2 and 5 years
  Change in the 10-word test from Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) between baseline and follow ups.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Jern, MD, PhD, Principal Investigator — Inst. of Biomedicine, the Sahlgrenska Academy, Univ. of Gothenburg; Turgut Tatlisumak, MD, PhD, Principal Investigator — Dept. of Neurology, Sahlgrenska Univ. Hosp., Gothenburg; Katarina Jood, MD, PhD, Principal Investigator — Dept. of Neurology, Sahlgrenska Univ. Hosp., Gothenburg
Locations (1):
- Department of Neurology, Department of Neurorehabilitation and Department of Clinical Genetics, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
Anonymized data may be shared by qualified academic research collaborators as long as data transfer is in agreement with EU legislation on the general data protection regulation and decisions by the Ethical Review Board of Sweden and the University of Gothenburg, which should be regulated in a data transfer agreement.

REFERENCES:
- [Background] Wieloch T, Nikolich K. Mechanisms of neural plasticity following brain injury. Curr Opin Neurobiol. 2006 Jun;16(3):258-64. doi: 10.1016/j.conb.2006.05.011. Epub 2006 May 18. PMID 16713245
- [Background] Doll DN, Barr TL, Simpkins JW. Cytokines: their role in stroke and potential use as biomarkers and therapeutic targets. Aging Dis. 2014 Oct 1;5(5):294-306. doi: 10.14336/AD.2014.0500294. eCollection 2014 Oct. PMID 25276489
- [Derived] Brannmark C, Klasson S, Stanne TM, Samuelsson H, Alt Murphy M, Sunnerhagen KS, Aberg ND, Jalnefjord O, Bjorkman-Burtscher I, Jood K, Tatlisumak T, Jern C. FIND Stroke Recovery Study (FIND): rationale and protocol for a longitudinal observational cohort study of trajectories of recovery and biomarkers poststroke. BMJ Open. 2023 May 10;13(5):e072493. doi: 10.1136/bmjopen-2023-072493. PMID 37164469